CLINICAL TRIAL: NCT00507663
Title: Elder Surgery - Functional Recovery Following Beta Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 00-0100; AG018772 (Other Grant/Funding Number: National Institute on Aging (NIA))
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Post Operative Cognitive Dysfunction
Keywords: beta blocker; functional recovery
MeSH Terms: interventions — Atenolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atenolol (Experimental): Atenolol given prior to and for up to 7 days after surgery
  Interventions: Drug: Atenolol
- routine care (No Intervention): routine clinical care

INTERVENTIONS:
Drug: Atenolol — Patients with a standing prescription for β-blockers will be continued on that medication. Pts not currently receiving a beta blocker will be given 50mg of atenolol on the morning of surgery, 50-100mg, twice per day, on the first postoperative day until postoperative day 7.
  Other Names: Tenormin
  Arms: Atenolol

SUMMARY:
This study proposes a prospective randomized study of elders undergoing elective major abdominal surgery to assess recovery following a unique anesthetic regimen incorporating a adrenergic receptor antagonist. The purposes of this study are to:

1. to determine if using atenolol, a beta-blocker drug commonly used to treat high blood pressure and heart disease, as part of your anesthetic regimen will decrease complications that sometimes occur in elderly patients who are undergoing surgery and being given anesthesia.
2. to see if it improves or quickens your recovery from anesthesia and surgery.
3. to help investigators design better ways to administer anesthesia during surgery, especially in elderly patients, so that the complications and the time to recover from surgery and anesthesia can be decreased.

DETAILED DESCRIPTION:
Increasing numbers of aged patients with multiple chronic diseases are undergoing major surgery. In the first third the last century, surgery was considered a desperate measure and patients greater than 50 years of age were felt incapable of sustaining the rigors of an inguinal hernia repair. Advances in anesthesia during the last century have allowed surgeons to develop an extraordinary array of procedures with excellent outcomes. Over 5.5 million patients aged 60 and over had major procedures in 1994. Centenarians routinely undergo surgical procedures.

Notwithstanding the enthusiasm for surgical treatments, morbidity, mortality, and recovery times for elderly patients are still substantially greater than for younger patients. Some morbidities, such as postoperative delirium and cognitive dysfunction appear to predominantly affect elderly patients. In a previous study, Dr. Valerie Lawrence, a co-investigator on this proposal, demonstrated that recovery from major surgery, as measured by the ability to accomplish standard activities of daily living, takes an average of 6 weeks while more complicated instrumental activities of daily living take an average of 3 months to return to baseline in elderly surgical patients. These data have profound implications for initiatives to control length of hospital stay, utilization of resources and costs of care. Evidence suggests that family members are requiring extra time off work to care for family members discharged earlier from hospitals.

Published reports and our preliminary data support the notion that intraoperative administration of adrenergic receptor antagonists (blockers) will improve functional recovery following surgery under general anesthesia. There is value in targeting functional status for elders undergoing surgery, because there is a direct relationship between functional status and utilization of health resources. Maximizing postoperative recovery, as opposed to minimizing morbidity and mortality, associated with surgical interventions in the elderly is consistent with the goal of prolonging "active life expectancy" expounded by Healthy People 2002.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years of age or older
* Patients undergoing elective major abdominal surgery (including but not limited to bowel, gastric, esophageal, pancreatic, gynecologic, urologic, and major intra-abdominal vascular procedures).
* Procedures requiring general anesthesia
* Laparoscopic-assisted major abdominal procedures
* Procedures requiring a 2-3 day postoperative stay will be included.

Exclusion Criteria:

* Unable to give informed consent to participate
* Folstein Mini-Mental State Examination Score < 17
* Gastrostomy tube placement
* Laparoscopic cholecystectomy, laparoscopic Nissen fundoplication, or any type of Hernia repair
* Appendectomy
* Emergency surgery
* Contraindications to adrenergic antagonists (third-degree heart block, decompensated congestive heart failure, active bronchospasm)
* Surgery within the previous month
* Major systemic infections
* Allergies to or incompatibilities with any drug used in this study
* Principle language other than English or Spanish
* Residence greater than 100 miles away from Manhattan
* Chronic debilitated state from which significant functional improvement following surgery is not anticipated (e.g., some nursing home residents, known metastatic cancer with poor prognosis)
* Chronic opioid usage
* Immunosuppression (subsequent opportunistic infections may obscure postoperative recovery).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 359 (Actual)
Dates: Start 2002-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Long Term Functional Recovery | at 3 weeks after surgery
  self reported Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL).

SECONDARY OUTCOMES:
Timed Up and Go test | preoperatively
  assesses basic functional mobility
Timed Up and Go test | once at 7-10 days postoperatively
  assesses basic functional mobility
Timed Up and Go test | 1 month postoperatively
  assesses basic functional mobility
Timed Up and Go test | 3 months postoperatively
  assesses basic functional mobility
Timed Up and Go test | 6 months postoperatively
  assesses basic functional mobility
Hand grip strength | preoperatively
  performance-based measure of upper extremity strength.
Hand grip strength | once at 7-10 days postoperatively
  performance-based measure of upper extremity strength.
Hand grip strength | 1 month postoperatively
  performance-based measure of upper extremity strength.
Hand grip strength | 3 months postoperatively
  performance-based measure of upper extremity strength.
Hand grip strength | 6 months postoperatively
  performance-based measure of upper extremity strength.

CONTACTS AND LOCATIONS:
Overall Officials: Jefrey H. Silverstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - The Mayo Clinic, Rochester, Minnesota
  - NYU School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York